CLINICAL TRIAL: NCT00077805
Title: An Open-Label, Randomized, Parallel-Group, Multi-Center Study to Evaluate the Efficacy and Safety of Enoxaparin Versus Unfractionated Heparin in the Prevention of Venous Thromboembolism in Patients Following Acute Ischemic Stroke
Brief Title: PREVAIL: PREvention of VTE After Acute Ischemic Stroke With LMWH Enoxaparin ( - VTE: Venous Thromboembolism - LMWH: Low Molecular Weight Heparin)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XRP4563H_4001
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — enoxaparin sodium

INTERVENTIONS:
Drug: Enoxaparin sodium

SUMMARY:
Primary objective:

* To demonstrate superiority of enoxaparin 40 mg sc qd in the prevention of VTE compared to UFH (unfractionated heparin) 5000 U sc q12 hours given for 10 ± 4 days following acute ischemic stroke.

Secondary objectives:

* To compare the incidence of VTE between the 2 treatment groups at 30, 60, and 90 days from the time of randomization
* To compare neurologic outcomes between the 2 treatment groups, including incidence of stroke recurrence, rate of stroke progression, and patient functional status, during the 10 ± 4 days of treatment, and after 30, 60, and 90 days from the time of randomization
* To evaluate the safety of using enoxaparin compared to UFH for VTE prevention in patients following acute ischemic stroke

ELIGIBILITY:
Inclusion criteria:

* Acute ischemic stroke, any territory, with an appropriate neuroradiologic study (head CT scan or brain MRI scan) providing results consistent with non hemorrhagic stroke
* Onset of symptoms of qualifying stroke within 48 hours prior to randomization. In patients receiving thrombolytic therapy for the acute stroke, such as tissue-type plasminogen activator (tPA), administration of study drug may not start until at least 24 hours after completion of thrombolytic therapy
* Significant motor impairment of the leg, as indicated by a NIHSS score ≥2 on item 6
* Inability to walk without assistance

Exclusion criteria:

* Females who are pregnant, breast-feeding, or of childbearing potential and not using medically acceptable and effective contraception
* Clinical evidence of VTE at screening
* Any evidence of active bleeding on the basis of clinical judgment
* Prior history of intracranial hemorrhage (including that at screening)
* Spinal or epidural analgesia or lumbar puncture within the preceding 24 hours
* Thrombolytic therapy (e.g., tPA) or intra-arterial thrombolytic therapy within the preceding 24 hours.Thrombolytic therapy is permitted for treatment of the acute stroke but must have been completed 24 hours prior to randomization.
* Comatose at screening (NIHSS score ≥2 on item 1a)
* Known or suspected cerebral aneurysm or arteriovenous malformation
* Confirmed malignancy that may pose an increased risk for bleeding or otherwise compromise follow-up or outcome assessment (e.g., lung cancer)
* Impaired hemostasis, i.e., known or suspected coagulopathy (acquired or inherited); baseline platelet count <100,000/mm3; aPTT 1.5 X the laboratory upper limit of normal; or international normalized ratio(INR) >1.5
* Major surgery or recent major trauma within the previous 3 months
* Anticipated need for full-dose treatment with therapeutic levels of an anticoagulant (LMWH, UFH, oral anticoagulant), e.g., for cardiogenic source of embolism or dissection
* Treatment with a LMWH or UFH at prophylactic dose for more than 48 hours prior to randomization(patients receiving LMWH or UFH less than 48 hours prior to randomization may be randomized)
* Allergy to heparin or enoxaparin sodium, or known hypersensitivity to heparin, enoxaparin, or pork products
* History of heparin or enoxaparin induced thrombocytopenia and/or thrombosis (heparin-induced thrombocytopenia [HIT], heparin-associated thrombocytopenia [HAT], or heparin-induced thrombotic thrombocytopenia syndrome [HITTS])
* History of hypersensitivity to iodinated contrast media and/or iodine
* Bacterial endocarditis
* Prosthetic heart valve
* Known or suspected severe anemia (Hg <10.0 g/dL)
* Uncontrolled arterial hypertension (systolic blood pressure [BP] >180 mmHg or diastolic BP >100 mmHg) at the time of randomization or clinical hypertensive urgency
* Any other clinically relevant serious diseases, including severe liver disease or renal failure [creatinine clearance <30 mL/min on at least two occasions].
* Treatment with other investigational agents or devices within the previous 30 days, planned use of other investigational drugs or devices, or previous enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Cumulative occurrence of VTE events (deep-vein thrombosis, pulmonary embolism) | 10 ± 4 days following acute ischemic stroke

SECONDARY OUTCOMES:
cumulative VTE events | at 30-day, 60-day and 90-day
stroke recurrence, stroke progression, National Institute of Health Stroke Scale (NIHSS) scores | during treatment and follow-up periods
Modified Rankin Scale (MRS) scores | at 30-day and 90-day follow-up
major & minor hemorrhages | from the inform consent signed up to the end of the study
Treatment emergent adverse events (TEAE), serious adverse events (SAE), all-cause mortality | from the inform consent signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Luc Sagnard, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, North Ryde, Australia
- Sanofi-Aventis, Vienna, Austria
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Bogotá, Colombia
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Mumbai, India
- Sanofi-Aventis, Netanya, Israel
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Johannesburg, South Africa
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Kase CS, Albers GW, Bladin C, Fieschi C, Gabbai AA, O'Riordan W, Pineo GF; PREVAIL Investigators. Neurological outcomes in patients with ischemic stroke receiving enoxaparin or heparin for venous thromboembolism prophylaxis: subanalysis of the Prevention of VTE after Acute Ischemic Stroke with LMWH (PREVAIL) study. Stroke. 2009 Nov;40(11):3532-40. doi: 10.1161/STROKEAHA.109.555003. Epub 2009 Aug 20. PMID 19696423
- [Result] Sherman DG, Albers GW, Bladin C, Fieschi C, Gabbai AA, Kase CS, O'Riordan W, Pineo GF; PREVAIL Investigators. The efficacy and safety of enoxaparin versus unfractionated heparin for the prevention of venous thromboembolism after acute ischaemic stroke (PREVAIL Study): an open-label randomised comparison. Lancet. 2007 Apr 21;369(9570):1347-1355. doi: 10.1016/S0140-6736(07)60633-3. PMID 17448820